CLINICAL TRIAL: NCT04836910
Title: The Change in Microbiome Following Treatment of Women With Polycystic Ovaries
Brief Title: Microbiome and Polycystic Ovaries
Status: Not yet recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Other Study IDs: 8032-20-SMC
Record Dates: First submitted 2021-03-25; First posted 2021-04-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Polycystic Ovary Syndrome; Microbial Colonization
Keywords: polycystic ovaries, microbiome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Communicable Diseases | interventions — World Health Organization; Metformin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples for microbiome analysis, vaginal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Women with Polycystic Ovary Syndrome: Woen diagnosed with Polycystic Ovary Syndrome according to the Rotterdam Criteria (requires 2 out of 3 symptoms: 1. Hyperandrogenism or excess levels of androgen. 2. Oligo or anovulation. 3. Polycystic ovaries on ultrasound - over 12 follicles, 2-9 mm or increased ovarian volume),who haven't started any treatment
  Interventions: Other: Dietary recommendations; Drug: Oral contraceptive pills; Drug: Metformin
- Cohort Group: Women without Polycystic Ovary Syndrome

INTERVENTIONS:
Other: Dietary recommendations — Fruit, vegetables, legumes (e.g. lentils and beans), nuts and whole grains (e.g. unprocessed maize, millet, oats, wheat and brown rice).
  At least 400 g (i.e. five portions) of fruit and vegetables per day excluding potatoes, sweet potatoes, cassava and other starchy roots.
  Less than 10% of total energy intake from free sugars Less than 30% of total energy intake from fats. Unsaturated fats (found in fish, avocado and nuts, and in sunflower, soybean, canola and olive oils) are preferable to saturated fats.
  Less than 5 g of salt (equivalent to about one teaspoon) per day.
  Other Names: World Health Organisation (WHO) recommendations
  Groups: Study Group: Women with Polycystic Ovary Syndrome
Drug: Oral contraceptive pills — Hormonal treatment
  Groups: Study Group: Women with Polycystic Ovary Syndrome
Drug: Metformin — Insulin resistance treatment
  Groups: Study Group: Women with Polycystic Ovary Syndrome

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is the most common endocrine disorder among women in reproductive age with an estimated prevalence of 5% to 19.5%. It is a chronic complex syndrome with psychological (depression and anxiety), reproductive and metabolic abnormalities. The etiology seems to be multifactorial. Lately, interest regarding the association between PCOS women and gut macrobiotic have been emerged. Hyperandrogenism was correlated with those changes in the microbiota which reflects the fact that the microbiome can influence the development and pathology of PCOS .

Therefore, aim of this study is to explore the diversity and alternations of the vaginal and the gut microbiome in patients with PCOS during common therapeutic interventions and connect them to different phenotypes of the syndrome.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is the most common endocrine disorder among women in reproductive age with an estimated prevalence of 5% to 19.5%. It is a chronic complex syndrome with psychological (depression and anxiety), reproductive and metabolic abnormalities. The etiology seems to be multifactorial. It seems there are both genetic, epigenetic and environmental contributors (almost 100 susceptible genes were identified).

The quality of life (QQL) of women suffering from PCOS is significantly reduced in all domains (functional ability, physical and emotional) and major health problems is correlated to PCOS. Women with PCOS demonstrate hyperinsulinemia and insulin resistance. They have an increased risk for type 2 diabetes and impaired glucose tolerance. Studies have shown that adipocyte function is considerably aberrant in women with PCOS including: lower lipase activity, defective glucose transport and dyslipidemia. Obesity is more prevalent in women with PCOS. They are also exposed to long term risk for additional disorders like cardiovascular diseases (atherosclerosis) or even cancer (endometrial or ovarian) .

PCOS is the primary cause of anovulatory subfertility. Furthermore, women with PCOS are at risk for pregnancy and obstetrical complications including preterm birth, pre- eclampsia and meconium aspiration syndrome of neonates after birth.

PCOS is diagnosed according the Rotterdam criteria . It requires 2 out of 3 symptoms: 1. Hyperandrogenism or excess levels of androgen)- clinical and/ or biochemical (presence of hirsutism, acne or alopecia). 2. Oligo or anovulation (including menstrual dysfunction). 3. PCO-M polycystic ovaries morphology (over 12 follicles, 2-9 mm or increased ovarian volume).

The term microbiome describes the genetic material of all the microbes (bacteria, fungi, protozoa and viruses) that live onside and inside the human body. It is important for development of the body, immunity and nutrition. The microbiome may influence the susceptibility to different infectious diseases and contribute to chronic illnesses.

The gut microbiota contains 100 trillion microbes. When discussing gut bacteria, it is primarily referred to the large intestine (colon). Lately, interest regarding the association between PCOS women and gut macrobiotic have been emerged. Hyperandrogenism was correlated with those changes in the microbiota which reflects the fact that the microbiome can influence the development and pathology of PCOS . Preliminary studies have shown that different bacterial species colonize the gut of PCOS induced animals compared to controls.

A novel theory was developed concerning the development of PCOS. A diet high of sugars sets as a convenient platform for gram negative bacteria ("bad" bacteria) while reducing "good" bacteria. The cell wall of the gram negative bacteria is comprised of lipopolysaccharide (LPS) which stimulates the immune system. The high sugar diet increases the permeability of the gut ("leaky gut") leading to chronic inflammation which produces impaired insulin receptor function. The insulin facilitates an increase in the production of androgens by the ovaries which leads to PCOS .

The dysbiosis was correlated with sex hormone levels and ovarian changes. In addition, treating PCOS using lactobacillus ("good" bacteria) transplantation showed improved ovarian functions.

Even though, several studies established the connection between the dysbiosis of the gut and PCOS, only a few studies were conducted on the association between the vaginal microbiome and the development of PCOS. To detail, the vaginal microbiome in PCOS is more diverse and heterogeneous, with the relative abundance of certain species (such as Mycoplasma) and lower level of others (such as Lactobacillus which keeps the vagina acidic) .

Moreover, should this association be strengthen between the microbiome of the gut and vagina to PCOS, it could serve as grounds to new horizons for treatment. There are several therapies for PCOS treatment (Life style interventions, improving metabolic dysfunction and medical treatment ), however, currently, there is no ideal therapy that fully treats all the clinical features.

Due to all the aforementioned, we aim of this study is to explore the diversity and alternations of the vaginal and the gut microbiome in patients with PCOS during common therapeutic interventions and connect them to different phenotypes of the syndrome.

Study design A prospective longitudinal case control study that will be conducted at Sheba Medical Center (tertiary medical center).

Study group will include 20 women in fertility age (age 18-42) diagnosed with PCOS according to the Rotterdam Criteria who haven't started any kind of treatment. The control group would be healthy women matched by age. Women in both groups will be recruited at the Endocrine outpatient's clinics. All women will sign informed consent form after receiving information on the study from one of the research team members.

Vaginal and rectal samples will be collected during the regular clinic visits that will be set by the medical interventions requirements (including: dietary recommendations, physical activity, hormonal contraception, insulin resistance treatment, fertility treatment, pregnancy follow-up):

1. at first visit after recruitment
2. 1 month following first intervention
3. 3 month following first intervention

ELIGIBILITY:
Inclusion Criteria:

Study group: Untreated women diagnosed with PCOS that are planned for intervention.

Control group: Women without PCOS visiting the gynecologic outpatient's clinics.

Exclusion Criteria:

1. Endocrine abnormality ( Cushing's syndrome, congenital adrenal hyperplasia, thyroid disorder, hyperprolactinemia and androgen-secreting tumor).
2. Premature ovarian failure 2. Active malignancy 3. Participants taking antibiotics/ probiotics, hormonal, vaginal or laxative medicine (in the previous week).

4. Vaginitis/ Pelvic Inflammatory Disease (PID)

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Study group will include 20 women in fertility age (age 18-42) diagnosed with PCOS according to the Rotterdam Criteria who haven't started any treatment. The control group would include healthy women matched by age.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Vaginal and gut microbiota composition before and after intervention recommended and in comparison to women without PCOS. | Through study completion, an estimated period of 1 year
  Evaluated by PCR ( ng/microl)

SECONDARY OUTCOMES:
Hirsutism | Through study completion, an estimated period of 1 year
  Change in hirsutism - subjectively reported by the women during clinic visits, on scale 0-4 (0-no change, 4-substantial improvement), and additionally evaluated before and after treatment by the Modified Ferriman-Gallwey Scoring (evaluating 9 body areas to assess hair growth (on 0-4 scale: 0-no hair growth to 4- extensive hair growth)
Acne | Through study completion, an estimated period of 1 year
  Change in Acne sevirity - subjectively reported by the women during clinic visits - Mild/ Moderate /Severe
Fertility | Through study completion, an estimated period of 1 year
  Sucess achieving pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Gynecology. ACOG Practice Bulletin No. 194: Polycystic Ovary Syndrome. Obstet Gynecol. 2018 Jun;131(6):e157-e171. doi: 10.1097/AOG.0000000000002656. PMID 29794677
- [Background] Macut D, Bjekic-Macut J, Rahelic D, Doknic M. Insulin and the polycystic ovary syndrome. Diabetes Res Clin Pract. 2017 Aug;130:163-170. doi: 10.1016/j.diabres.2017.06.011. Epub 2017 Jun 12. PMID 28646699
- [Background] Lizneva D, Suturina L, Walker W, Brakta S, Gavrilova-Jordan L, Azziz R. Criteria, prevalence, and phenotypes of polycystic ovary syndrome. Fertil Steril. 2016 Jul;106(1):6-15. doi: 10.1016/j.fertnstert.2016.05.003. Epub 2016 May 24. PMID 27233760
- [Background] McCartney CR, Marshall JC. CLINICAL PRACTICE. Polycystic Ovary Syndrome. N Engl J Med. 2016 Jul 7;375(1):54-64. doi: 10.1056/NEJMcp1514916. PMID 27406348
- [Background] Azziz R. Polycystic Ovary Syndrome. Obstet Gynecol. 2018 Aug;132(2):321-336. doi: 10.1097/AOG.0000000000002698. PMID 29995717
- [Background] Azziz R, Carmina E, Chen Z, Dunaif A, Laven JS, Legro RS, Lizneva D, Natterson-Horowtiz B, Teede HJ, Yildiz BO. Polycystic ovary syndrome. Nat Rev Dis Primers. 2016 Aug 11;2:16057. doi: 10.1038/nrdp.2016.57. PMID 27510637
- [Background] Lindheim L, Bashir M, Munzker J, Trummer C, Zachhuber V, Leber B, Horvath A, Pieber TR, Gorkiewicz G, Stadlbauer V, Obermayer-Pietsch B. Alterations in Gut Microbiome Composition and Barrier Function Are Associated with Reproductive and Metabolic Defects in Women with Polycystic Ovary Syndrome (PCOS): A Pilot Study. PLoS One. 2017 Jan 3;12(1):e0168390. doi: 10.1371/journal.pone.0168390. eCollection 2017. PMID 28045919
- [Background] Hong X, Qin P, Huang K, Ding X, Ma J, Xuan Y, Zhu X, Peng D, Wang B. Association between polycystic ovary syndrome and the vaginal microbiome: A case-control study. Clin Endocrinol (Oxf). 2020 Jul;93(1):52-60. doi: 10.1111/cen.14198. Epub 2020 May 7. PMID 32311120